CLINICAL TRIAL: NCT07084909
Title: Phase 2/3 Open-Label Multicenter Study to Assess the Diagnostic Performance of Piflufolastat F 18 PET/CT on Intended Clinical Management in Patients With Suspected, or at High Risk for Metastatic ccRCC
Brief Title: Piflufolastat F 18 PET/CT in Patients With Suspected, or at High Risk for Metastatic ccRCC
Acronym: HARRIER
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Operational challenges in patient enrollment
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PYL2302
Record Dates: First submitted 2025-05-30; First posted 2025-07-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: kidney cancer; renal cell carcinoma; clear cell; Piflufolastat F 18; PYLARIFY; imaging; ccRCC; PET/CT
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2 - Dose Optimization (Experimental): The dose-optimization, or Phase 2, part of the study will enroll 6-12 ccRCC patients, with at least one metastatic lesion identified by conventional imaging at the time of enrollment, to define the optimal dose and scan timing window for piflufolastat F18 PET/CT. Piflufolastat F18 will be administered at a target dose of 9 mCi [+/-1 mCi]) after which patients will be scanned at 60-90 minutes and again at 3-4 hours.
  Interventions: Drug: piflufolastat F 18
- Phase 3 - Single-arm Expansion (Experimental): Phase 3 will commence once the optimal dose and optimal timing window from Phase 2, dose optimization, are determined. Phase 3 will be a single-arm study that will enroll 274 patients with radiographically suspected metastatic disease by conventional imaging or at high risk for metastatic ccRCC at the time of enrollment.
  Interventions: Drug: piflufolastat F 18

INTERVENTIONS:
Drug: piflufolastat F 18 — 18F-DCFPyL is a fluorine-18 radiolabeled low molecular weight positron emission tomography (PET) tracer that binds to the extracellular domain of prostate-specific membrane antigen (PSMA) with high affinity.
  Other Names: PYLARIFY

SUMMARY:
This study is being conducted to test whether an imaging technique called a "piflufolastat F 18 PET/CT" imaging scan can be used to diagnose and describe the extent of clear cell Renal Carcinoma in patients.

The main questions it aims to answer are:

* What is the most appropriate dose and scan timing window for piflufolastat F 18 PET/CT for patients with clear cell Renal Cell Carcinoma (ccRCC) with known metastatic disease?
* Ability of piflufolastat F 18 PET/CT to detect metastatic of lesions ccRCC in patients with suspected metastatic disease and those at high risk for metastatic disease (the cancer has spread beyond the kidney) and impact of the imaging on clinical management of the kidney cancer?

Participants will:

* Receive a single injection of piflufolastat F 18 injection followed by imaging scans.
* Be contacted via telephone to ask about any reactions or discomforts they may have after the piflufolastat F 18 injection.
* May be followed for up to 6 months to collect data about disease progression.

DETAILED DESCRIPTION:
This is an adaptive Phase 2/3, open-label, multi-center, single-arm study designed to evaluate diagnostic performance of piflufolastat F 18 PET/CT in the staging of patients suspected of having, or who are at high risk for, metastatic ccRCC and its impact on intended clinical management.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age
2. Patients must have the ability to understand and sign an approved informed consent form (ICF)
3. Patients must have the ability to understand and comply with all protocol requirements.
4. Subjects should satisfy the following criteria:

1) For the Phase 2 (dose optimization) portion of the study: ccRCC patients with at least one suspected metastatic lesion identified by conventional imaging scans at the time of enrolling in the study 2) For the Phase 3 portion of the study: Patients must be suspected of having or be at high risk for developing metastatic disease. This patient population is generally defined as one of the following:

1. Newly diagnosed ccRCC patients or post- nephrectomy/post-partial nephrectomy patients with radiographically suspected ccRCC metastatic disease by conventional imaging (CI) planned for biopsy to confirm metastatic disease
2. T2B-T4, N0, M0 as assessed by conventional imaging (CI) at initial staging pre-nephrectomy/pre-partial nephrectomy
3. Confirmed ccRCC with high risk of metastatic recurrence post nephrectomy pT1b or higher with G3-4 N0( or pNX where clinically N0)M0. Patients must be N0, M0 on the follow up CI not more than 60 days prior to piflufolastat F18 scan
4. Patients with new radiographically suspected oligometastatic ccRCC (up to 5 metastatic lesions at presentation) planned for nephrectomy or biopsy for lesion verification of at least one suspected metastatic lesion

   5. Completed staging evaluation with baseline conventional imaging (contrast-enhanced CT or contrast-enhanced MRI of the chest, abdomen, and pelvis, or skull base to mid thigh FDG PET)less than or equal to 60 days prior to piflufolastat F 18 PET/CT (Day 1). If baseline conventional imaging was performed outside of the 60-day window, it can be repeated during the screening period provided that there are at least 24 hours between conventional imaging and piflufolastat F 18 (Day 1). Conventional imaging must be available for central evaluation.

   6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

   7. Patients with life expectancy of at least 6 months as determined by the investigator or treating physician.

   Exclusion Criteria:
   1. Patients administered any high energy (>300 KeV) gamma-emitting radioisotope within five (5) physical half-lives, prior to Day 1.
   2. Known hypersensitivity to the components of piflufolastat F 18 or its analogs.
   3. Pregnant or breastfeeding females. Pregnancy testing will be performed in potentially childbearing women prior to piflufolastat F 18 administration on Day 1.
   4. Prior imaging with girentuximab or any PSMA-PET agent or any non-approved ccRCC imaging agent within the last 3-months prior to piflufolastat F 18 PET/CT.
   5. Patients who are in active systemic therapy for metastatic ccRCC prior to piflufolastat F 18 PET/CT. 30-day (12 weeks for immunotherapy) washout period is required from the last dose of systemic therapy to piflufolastat F18 administration.
   6. Patients who are expected to receive anti-cancer treatment between baseline conventional imaging, piflufolastat F 18 PET/CT, biopsy, or surgery.
   7. Evidence of any other active malignancy within the past 3 years, except non-melanoma skin cancer, carcinoma in situ, adequately treated Stage 1 cancer from which the patent is in remission and has been in remission for a minimum of 2 years. Any adjuvant or maintenance systemic chemotherapy must have been completed at least 30 days prior to piflufolastat F 18 PET/CT administration (12-week washout if immunotherapy).
   8. Patients with any medical condition or other circumstances that, in the opinion of the investigator, compromise the safety or compliance of the subject to produce reliable data or completing the study.
   9. Patients requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Phase 2 Primary Objective - Establishing the optimum dose and timing window of piflufolastat F18 for detection of metastatic disease | On Day 1 (day of injection) where Piflufolastat F18 will be administered at a target dose of 9 mCi [+/-1 mCi]) after which patients will be scanned at 60-90 minutes and again at 3-4 hours.
  Defining the optimal dose and scan timing window for Piflufolastat F18 PET/CT
Phase 3 Primary Objective - To assess the diagnostic performance of piflufolastat F 18 PET/CT to determine the presence or absence of metastatic disease in ccRCC patients. | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration to establish the standard of truth.
  Sensitivity of piflufolastat F 18 PET/CT at the patient level to determine the presence of metastatic ccRCC relative to the composite truth standard. Specificity of piflufolastat F 18 PET/CT at the patient level to determine the absence of metastatic ccRCC relative to the composite truth standard.

SECONDARY OUTCOMES:
Phase 3 -To assess the diagnostic performance of piflufolastat F 18 PET/CT for identifying the presence of metastatic lesions in ccRCC | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration to establish the standard of truth.
  Correct localization rate (CLR) at the patient level, defined as the percentage of patients for whom there is a one-to-one correspondence between localization of at least one lesion identified on piflufolastat F 18 PET CT and a composite standard of truth (SOT)
Phase 3 - Safety and Tolerability | From screening to to 6 months post-piflufolastat F 18 administration
  Incidence of adverse events (AEs), changes in vital signs, clinical laboratory parameters and concomitant medications.
Phase 3 - Assess the impact of piflufolastat F 18 PET/CT on intended and actual patient clinical management | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration
  Change in intended and actual patient clinical management in all patients as assessed by a Medical Management Questionnaire (MMQ)

OTHER OUTCOMES:
Exploratory - Assess the sensitivity of piflufolastat F 18 PET/CT at the Lesion Level | From screening to 6 months post-piflufolastat F 18 administration
  Sensitivity of piflufolastat F 18 PET/CT at the lesion level to determine the presence of metastatic ccRCC relative to the composite truth standard, if possible
Exploratory - Measure PSMA expression and neovascular localization in metastatic lesions using immunohistochemistry (IHC) | At 3 months and 6 months post-piflufolastat F 18 administration
  Use of IHC to assess PSMA expression and neovascular localization. Biopsy and surgery specimens obtained during the SOT follow-up period post PSMA PET will be analyzed for histopathology at the local laboratory, and for PSMA expression by IHC at a central laboratory.
Exploratory - Correlate circulating tumor DNA (ctDNA) levels and tumor specific genetic signatures with tumor burden assessed by piflufolastat F 18 PET imaging and PSMA IHC | At the time surgical/biopsy samples are obtained
  ctDNA sequencing will be performed to assess ctDNA levels and tumor-specific genetic signatures which may be correlated with piflufolastat F 18 PET/CT and PSMA IHC
Exploratory - Compare piflufolastat F 18 PET/CT findings with PSMA expression levels in metastatic lesions as assessed using IHC | Prior to piflufolastat F 18 dosing through surgical/biopsy sampling
  Correlation of piflufolastat F 18 uptake parameters (including, but not limited to SUV peak, SUV mean, SUV max) and PSMA expression levels in metastatic lesions determined by IHC will be calculated.
Exploratory - To Determine Positive Predictive Value (PPV) | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration
  Positive Predictive Value (PPV) of piflufolastat F 18 PET/CT in the detection of metastatic ccRCC at a lesion level
Exploratory - utility of aPROMISE in patients with metastatic ccRCC | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration
  PSMA score, number of lesions, and SUV values will be calculated using aPROMISE to generate quantification of disease burden in patients with metastatic ccRCC
Exploratory - Compare aPROMISE assessment with PSMA expression | From Day 1 (day of injection) where Piflufolastat F18 will be administered to 6 months post-piflufolastat F 18 administration
  Correlation of aPROMISE results and PSMA expression in metastatic lesions assessed using IHC

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - XCancer, Omaha, Nebraska